CLINICAL TRIAL: NCT01488773
Title: A Four Year Observational Study Comparing Two Treatment Regimens: Inhaled Glucocorticosteroid + Salmeterol and Inhaled Glucocorticosteroid + Montelukast.
Brief Title: Comparison of Two Treatment Regimens in Asthmatic Patients
Status: Completed | Type: Observational
Sponsor: Medical University of Lodz (Other)
Responsible Party: Principal Investigator, Rafal Pawliczak, MD PhD, Prof. Rafal Pawliczak, Medical University of Lodz
Other Study IDs: adamusiak-01
Record Dates: First submitted 2011-12-06; First posted 2011-12-08 (Estimated); Last update posted 2012-01-12 (Estimated); Status verified 2012-01

CONDITIONS: Asthma
Keywords: asthma; asthma control; inhaled glucocorticosteroid; ICS; leukotriene antagonist; LTRA; montelukast; fluticasone; salmeterol; observational study; repeated measures; retrospective
MeSH Terms: conditions — Asthma | interventions — montelukast; Salmeterol Xinafoate

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- ICS + salmeterol: Patients treated with both inhaled glucocorticosteroid (ICS) and salmeterol (long-acting β2-agonist).
  90 patients met the inclusion criteria for this group.
  Interventions: Drug: first prescription of salmeterol
- ICS + montelukast: Patients treated with both inhaled glucocorticosteroid (ICS) and montelukast (leukotriene receptor antagonist).
  42 patients met the inclusion criteria for this group.
  Interventions: Drug: first prescription of montelukast

INTERVENTIONS:
Drug: first prescription of montelukast — The index event (intervention) was defined as the first prescription for montekuast (leukotriene receptor antagonist) occurring in patient's medical history that established a 12-month pre-index and three consecutive 12-month post-index periods.
  Other Names: Singulair
  Groups: ICS + montelukast
Drug: first prescription of salmeterol — The index event (intervention) was defined as the first prescription for salmeterol (long-acting β2-agonist) occurring in patient's medical history that established a 12-month pre-index and three consecutive 12-month post-index periods.
  Other Names: Serevent
  Groups: ICS + salmeterol

SUMMARY:
The objective of the study was to compare in real life clinical practice two treatment regimens: inhaled glucocorticosteroid + salmeterol and inhaled glucocorticosteroid + montelukast.

DETAILED DESCRIPTION:
48 month pre/post retrospective repeated measures design was used to compare the level of asthma control among patients continuously treated at the Outpatient Asthma and Allergy Treatment Center, Chair of Clinical Immunology and Microbiology, Medical University of Lodz, Poland.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of asthma according to the WHO/GINA 2006 definition by the physicians of the Centre, backed up by detailed medical history and physical examination as well as additional spirometry and bronchodilatation test or methacholine challenge where necessary
* Occurrence of an index event (intervention) defined as the first prescription for salmeterol or montelukast, establishing a 12-month pre-index and three consecutive 12-month post-index periods
* At least one inhaled glucocorticosteroid prescription in the pre-index period, and at least one salmeterol/montelukast prescription depending on the arm in every post-index period

Exclusion Criteria:

* Incomplete diagnostics

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population consisted of 5563 patients continuously treated for bronchial asthma (28% of all patients) at the Outpatient Asthma and Allergy Treatment Center, Chair of Clinical Immunology and Microbiology, Medical University of Lodz, Poland in the period from April 1995 through June 2006.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 1995-04; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Asthma Control Index | 12 months
  A composite measure based on GINA 2006 guidelines and Asthma Control Questionnaire© (ACQ) by Juniper et al. Each of the five parameter was assessed on a three-level scale 2 - 1 - 0 and summed up to provide the final score between 0 (uncontrolled asthma) and 10 (controlled asthma). These parameters were:
  Nocturnal dyspnea (none, 1, 1+);Daytime dyspena (none, 1, 1+);Wheeze (none, 1, 1+);short-acting β2-agonist utilization (0, less or half a container a year, more than half a container a year);FEV1 (>90%,>80%,<80%)

SECONDARY OUTCOMES:
number of outpatient visits | 12 months
number of asthma-related hospitalizations | 12 months
mean value of pulmonary function tests (PEF and FEV1) | 12 months
number of doctor-defined asthma exacerbations | 12 months
number of acute respiratory infections | 12 months
number of nocturnal and day-time dyspneas | 12 months
number of episodes of wheeze | 12 months
exact prescribed doses of anti-inflammatory drugs | 12 months
number of prescribed containers of short-acting β2-agonists, antihistamines, and antibiotics | 12 months
number of pulmonary function tests declines below 80% personal best | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Rafal Pawliczak, MD PhD, Principal Investigator — Department of Immunopathology Chair of Allergy, Immunology and Dermatology Faculty of Biomedical Sciences and Postgraduate Training Medical University of Lodz